CLINICAL TRIAL: NCT06855355
Title: Clostridium Butyricum MIYAIRI 588 Reduces Colorectal Adenomatous Polyp Recurrence: A Randomized Crossover Trial
Brief Title: CBM588 Reduces Colorectal Polyp Recurrence
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Jiunn-Wei Wang, Doctor, Kaohsiung Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CBM588 and Colorectal Polyp
Record Dates: First submitted 2025-02-11; First posted 2025-03-03 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Polyp
Keywords: gut microbiota; butyrate-producing bacteria; probiotic therapy; colorectal neoplasia prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBM588 First-Year Treatment Group (Group A) (Experimental): .Participants receive Clostridium butyricum MIYAIRI 588 (CBM588) for one year. .Followed by a washout period and no treatment in the second year. .Annual colonoscopies are performed to assess polyp recurrence.
  Interventions: Dietary Supplement: Clostridium butyricum MIYAIRI 588
- CBM588 Second-Year Treatment Group (Group B) (Active Comparator): .Participants do not receive CBM588 in the first year. .Undergo a washout period and then begin CBM588 treatment in the second year. .Annual colonoscopies are performed to assess polyp recurrence.
  Interventions: Dietary Supplement: Clostridium butyricum MIYAIRI 588

INTERVENTIONS:
Dietary Supplement: Clostridium butyricum MIYAIRI 588 — A butyrate-producing probiotic, has demonstrated potential anti-inflammatory and anti-tumorigenic effects.
  Other Names: MIYARISAN BM

SUMMARY:
The goal of this randomized crossover clinical trial is to evaluate the efficacy of Clostridium butyricum MIYAIRI 588 (CBM588) in reducing colorectal adenomatous polyp recurrence in adult patients with a history of colorectal polyps.

The main questions it aims to answer are:

* Does CBM588 reduce the recurrence of colorectal adenomatous polyps?
* Does CBM588 lead to a sustained decrease in polyp burden over time? Researchers will compare a group receiving CBM588 in the first year to a group receiving CBM588 in the second year (after a washout period) to determine whether CBM588 effectively lowers polyp recurrence rates and adenoma prevalence.

DETAILED DESCRIPTION:
This randomized crossover clinical trial evaluates the effect of Clostridium butyricum MIYAIRI 588 (CBM588), a butyrate-producing probiotic, on colorectal adenomatous polyp recurrence. Participants who had undergone complete polypectomy were randomly assigned into two groups:

* Group A: Received CBM588 for one year, followed by a washout period and no treatment in the second year.
* Group B: Did not receive CBM588 in the first year but received it in the second year after a washout period.

Annual colonoscopy assessments were conducted to evaluate polyp count, type, and location. The primary outcome measure is adenoma recurrence. This study was conducted at a tertiary medical center and received Institutional Review Board (IRB) approval (KMUHIRB-F(I)-20170010). All participants provided informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a history of colorectal adenomas that had been completely removed by endoscopic resection within the past three years, and who presented with recurrent colorectal polyps detected during surveillance colonoscopy
* Willingness to undergo follow-up colonoscopies at study intervals
* No antibiotic or probiotic use for at least three months before study entry
* Written informed consent obtained

Exclusion Criteria:

* History of colorectal cancer or other gastrointestinal malignancies
* Diagnosis of inflammatory bowel disease or familial adenomatous polyposis
* Use of antibiotics and other probiotics during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Colorectal polyp recurrence rate (%) | 1 year and 2.25 years after baseline colonoscopy
  The percentage of participants with at least one recurrent colorectal polyp detected during follow-up colonoscopy. Recurrence is defined as the presence of new polyps (adenomatous or non-adenomatous) identified on annual surveillance colonoscopy.

SECONDARY OUTCOMES:
Adenomatous polyp recurrence rate (%) | 1 year and 2.25 years after baseline colonoscopy
  The percentage of participants with at least one recurrent adenomatous polyp detected during follow-up colonoscopy.
Mean number of recurrent polyps | 1 year and 2.25 years after baseline colonoscopy
  The average number of polyps detected per participant during follow-up colonoscopy.
Polyp location distribution | 1 year and 2.25 years after baseline colonoscopy
  The proportion of recurrent polyps found in different segments of the colon (right colon, left colon, rectum).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) from this study. The primary reasons include privacy concerns, ethical considerations, and regulatory restrictions. The data contain sensitive health information, and sharing could compromise participant confidentiality. Additionally, there are no institutional or legal frameworks in place to support external data sharing for this study.